CLINICAL TRIAL: NCT03155373
Title: The Right Ventricular Pulmonary Circulation Continuum in Mitral Valve Disease
Brief Title: The Right Ventricular Pulmonary Circulation Continuum in Mitral Valve Disease Study
Acronym: RIPCOM1
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 16HH3639; 16/LO/2127 (Other: REC); 199676 (Other: IRAS)
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Mitral Regurgitation; Pulmonary Hypertension
Keywords: Cardiopulmonary exercise testing
MeSH Terms: conditions — Mitral Valve Insufficiency; Hypertension, Pulmonary | interventions — Cardiac Catheterization; Exercise Test; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Left and right ventricular biopsies taken at time of clinically indicated surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A: Asymptomatic/mild symptomatic patients with normal pre-operative left ventricular function (defined as left ventricular ejection fraction >60%)
  Interventions: Diagnostic Test: Cardiac catheterisation; Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: Pulmonary function tests; Diagnostic Test: Cardiac MRI; Other: Quality of life survey; Procedure: Mitral valve operation; Procedure: Myocardial biopsies
- B: Symptomatic patients with normal pre-operative left ventricular function (defined as left ventricular ejection fraction greater than or equal to 60%)
  Interventions: Diagnostic Test: Cardiac catheterisation; Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: Pulmonary function tests; Diagnostic Test: Cardiac MRI; Other: Quality of life survey; Procedure: Mitral valve operation; Procedure: Myocardial biopsies
- C: Patients with impaired pre-operative left ventricular function (defined as left ventricular ejection fraction <60%)
  Interventions: Diagnostic Test: Cardiac catheterisation; Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: Pulmonary function tests; Diagnostic Test: Cardiac MRI; Other: Quality of life survey; Procedure: Mitral valve operation; Procedure: Myocardial biopsies

INTERVENTIONS:
Diagnostic Test: Cardiac catheterisation — Pre-operative left heart catheterisation +/- right heart catheterisation
Diagnostic Test: Cardiopulmonary exercise testing — Pre and post-operative cardiopulmonary exercise testing
Diagnostic Test: Pulmonary function tests — Pre and post-operative pulmonary function tests
Diagnostic Test: Cardiac MRI — Pre and post-operative cardiac MRI
Other: Quality of life survey — Pre and post-operative quality of life survey (SF36)
Procedure: Mitral valve operation — Clinically indicated mitral valve repair/replacement +/- coronary artery surgery +/- tricuspid valve surgery +/- atrial fibrillation surgery
Procedure: Myocardial biopsies — Right and left epicardial ventricular biopsies taken at time of clinically indicated surgery

SUMMARY:
Mitral regurgitation (MR) is a prevalent valvular heart pathology. Indications for surgery include symptoms, impaired left ventricular function or enlarging dimensions, new onset atrial fibrillation, pulmonary hypertension, asymptomatic status with a high likelihood of success.

Asymptomatic severe primary MR can be initially monitored without impairing long term survival. However, significant symptoms or impairment of left ventricular function is associated with worse prognosis due to long term heart failure. Some physicians wait for early symptoms before referring for surgery and this is reflected by a great variation in referral patterns, but symptomatic status is subjective and difficult to assess. Nearly all of the surgical indications are based on expert opinion rather than significant evidence base.

The primary aim of this project is to improve the current guidelines for surgery for primary MR by finding an objective marker of functional capacity which correlates with surrogates of prognosis and detects early decline, but returns to normal after surgery.

DETAILED DESCRIPTION:
The current indications for surgery for MR include symptomatic status; asymptomatic status with echocardiographic features such as impaired left ventricular function or increased left ventricular dimensions; new onset atrial fibrillation or pulmonary hypertension; asymptomatic status with a high likelihood of durable repair and low co-morbidity. The limitation in strength of the current evidence base is reflected by the class of evidence being expert opinion (level C) for all of the above indications with the sole exception of symptomatic patients, which is level B.

The fulcrum point between asymptomatic status and symptomatic status at which patients would derive prognostic benefit and thus should be referred for surgery on prognostic grounds still remains unclear and controversial. Although elective mitral valve repair carries a low risk of mortality, it has been demonstrated that asymptomatic patients with severe degenerative MR can be safely followed up before becoming symptomatic or reaching cutoff values for left ventricular dimensions, size or pulmonary hypertension; with no significant difference with expected survival. As a result, it is debatable whether prophylactic surgery for all patients with asymptomatic severe degenerative MR derives prognostic benefit.

At the other end of the clinical spectrum, the increased operative mortality and worse long term prognosis of symptomatic patients is well proven. Patients with New York Heart Association Class III or IV status have excessive operative mortality and significantly increased mortality at 10 years. Both this study and another have demonstrated that preoperative ejection fraction is an independent predictor of long term survival. Although this evidence base does not support prophylactic surgery on asymptomatic patients, it does highlight the importance of avoiding the long term sequelae of MR in causing symptomatic status or left ventricular impairment. Hence attention has turned to objective markers or investigations independent of symptomatic status that may be subjectively assessed in the early phases; to help identify patients who would prognostically benefit from earlier surgical intervention.

In summary, severe mitral regurgitation is a common valvular pathology that causes a significant burden of disease. Current guidelines for timing of operative intervention are mostly based on expert opinion rather than randomised trials or studies. The ideal tipping point investigation will be an objective marker of functional capacity which correlates with known surrogates of survival such as left ventricular function; and detects early decline, but returns to normal after successful surgery. The improved evidence base will create an epidemiological shift in patterns of referring for mitral valve surgery and reduce the burden of disease of heart failure.

Patients will undergo the following investigations:

Right heart catheterisation- It is the usual gold standard practice at our institution for patients to have a right heart catheterisation before being referred for surgery. Those who have not had one may be referred to the Department of Cardiology at Hammersmith Hospital for this test.

Cardiac MRI- patients will have a T1 weighted cardiac MRI. One strength of cardiac MRI over transthoracic echocardiogram is objective measurements of right heart function. Parameters measured will be ventricular ejection fraction and dimensions, patterns of myocardial fibrosis.

Cardiopulmonary exercise testing (CPEX)- CPEX is a quantitative and validated method of assessing cardiorespiratory function and exercise capacity with commonly measured variables including maximal oxygen consumption (VO2 max) and the clearance of carbon dioxide during exercise (Ve/VCO2). The patient's gaseous exchange is monitored during a 3 minute rest period, a three minute "rolling basal" period when they perform exercise on a bicycle with no load; and subsequently during the exercise phase when the work load increases at a rate of 30 Watts per minute. Exercise continues until the patient has to stop or achieves predicted maximum heart rate.

Pulmonary function tests- Patients will have routine spirometry tests and also assessment of transfer factor.

Transthoracic echocardiogram- It is normal practice for patients to have an echocardiogram at preassessment clinic to assess biventricular function, dimensions and cardiac structural disease.

Quality of life questionnaire- Patients will be asked to fill out a validated questionnaire (SF-36 health survey).

ELIGIBILITY:
Inclusion Criteria:

Patients listed for surgery for severe primary mitral regurgitation +/- concomitant coronary artery bypass grafting for bystander disease +/- tricuspid valve surgery +/- atrial fibrillation surgery.

Exclusion Criteria:

Secondary mitral regurgitation. Significant history of ischaemic heart disease eg. angina. Age <18 years or >85 years. Critical preoperative status with multi-organ dysfunction. Emergency cardiac surgical intervention. Pregnancy. Unable to give informed consent or unwilling to participate in research. Patients with definite contraindication for MRI would be excluded from the cardiac MRI element of the study.

Patients we are unable to take adequate biopsies due to technical difficulties would be excluded from the myocardial biopsy element of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery for severe primary/degenerative mitral regurgitation under the current guidelines.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Punjabi, FRCS, Principal Investigator — Imperial College London; Simon Gibbs, FRCP, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Cohort: Patients undergoing surgery under current guidelines for surgery for primary MR.
Period: Overall Study
Arm/Group | Overall Cohort
Started | 50
Completed | 43
Not Completed | 7
Not completed — No longer required surgery | 1
Not completed — Protocol Violation | 1
Not completed — Death | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Overall Cohort
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 43

OUTCOME MEASURES:

1. Primary Outcome: Impaired Post-operative Functional Capacity
Description: Dichotomic variable of post-operative left ventricular ejection < 50% and/or post-operative percentage predicted peak VO2 <= 84%
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Overall Cohort: Patients meeting current international guidelines indications for surgery for primary mitral regurgitation
  Cardiac catheterisation: Pre-operative left heart catheterisation +/- right heart catheterisation
  Cardiopulmonary exercise testing: Pre and post-operative cardiopulmonary exercise testing
  Pulmonary function tests: Pre and post-operative pulmonary function tests
  Cardiac MRI: Pre and post-operative cardiac MRI
  Quality of life survey: Pre and post-operative quality of life survey (SF36)
  Mitral valve operation: Clinically indicated mitral valve repair/replacement +/- coronary artery surgery +/- tricuspid valve surgery +/- atrial fibrillation surgery
  Myocardial biopsies: Right and left epicardial ventricular biopsies taken at time of clinically indicated surgery
Arm/Group | Overall Cohort
Number analyzed (Participants) | 43
Participants | 35

2. Primary Outcome: Imaging Data
Description: Correlation between transthoracic echocardiogram and cardiac MRI parameters
Time Frame: 1 year
Population: Correlation co-efficient on linear model between LVEF measurement on transthoracic echocardiogram against cardiac MRI
Measure: Number; unit: r value
Arm/Group | Overall Cohort
Number analyzed (Participants) | 43
r value | 0.31

3. Secondary Outcome: Right Heart Catheterisation
Description: Accuracy of measurements of pre-op pulmonary artery pressures against the gold standard of right heart catheterisation
Time Frame: Pre-op
Population: Data were not collected since right heart catheterisation was not performed due to adding an extra invasive investigation on the patients after they had already met the guidelines for surgery.
Arm/Group | Overall Cohort
Number analyzed (Participants) | 0

4. Secondary Outcome: Quality of Life as Assessed by SF36 Survey
Description: Changes in quality of life measured on the SF36 survey after surgery
Time Frame: Baseline (preoperatively), early follow up (6 weeks after surgery), late follow up (6 months after surgery)
Population: Physical functioning on SF36 quality of life questionnaire from 0 (worst) to 100 (best) at baseline (preoperatively), early follow up (6 weeks after surgery), late follow up (6 months after surgery)
Measure: Mean (Standard Deviation); unit: Score on the scale
Arm/Group | Overall Cohort
Number analyzed (Participants) | 43
Score on the scale
  Pre-operative | 64.3 (26.6)
  Early follow up | 62.9 (25.4)
  Late follow up | 74.9 (23.7)

5. Secondary Outcome: Myocardial Histology
Description: Quantification of myocardial fibrosis on right and left ventricular biopsies
Time Frame: At surgery
Population: 15 patients consented to myocardial biopsies at time of surgery
Measure: Mean (Standard Deviation); unit: % interstitial fibrosis
Arm/Group | Overall Cohort
Number analyzed (Participants) | 15
% interstitial fibrosis
  RV in peak VO2>80% | 8.9 (2.2)
  RV in peak VO2 <80% | 8.4 (4.2)
  LV in peak VO2 >80% | 3.7 (2.3)
  LV in peak VO2 <80% | 7.4 (5.3)

ADVERSE EVENTS:
Time Frame: Each participant was assessed for 2 years after surgery
Arm/Group | Overall Cohort
All-Cause Mortality (participants affected / at risk) | 2/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
In the initial planning of this project, there were 3 defined arms. However, due to the small n number of patients recruited; there were insufficient numbers for meaningful analysis. Professional statistical advice was to analyse the entire cohort with the pre-defined dichotomous outcome of impaired functional status based on current evidence base/international guidelines (post-op LVEF <50% and percentage predicted peak VO2 <=84%) and a multivariate analysis of four pre-defined variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-12-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT03155373/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT03155373/SAP_001.pdf